CLINICAL TRIAL: NCT07134062
Title: The Effect of the Bridge Technique Mobilization With Movement Versus Trapezius Dry Needling in the Management of Cervical Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 117/REC/2020
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2020-03

CONDITIONS: Mulligan Mobilization; Dry Needling Technique; Physical Therapy
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Bridge technique mobilization with movement (Active Comparator): Patient in supine, head resting on a pillow, cervical spine relaxed in a neutral position, physiotherapist sitting or standing at the head of the table. Hands support both sides of the head through the thenar eminence on each side, fingers in contact with the C7, T1or T2 articular pillar bilaterally
  Interventions: Other: Bridge technique MWM
- Group 2 Dry Needling (Active Comparator): Participants in this group received two sessions per week of D.N. treatment for the trapezius muscle.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Bridge technique MWM — Patient in supine, head resting on a pillow, cervical spine relaxed in a neutral position, physiotherapist sitting or standing at the head of the table. Hands support both sides of the head through the thenar eminence on each side, fingers in contact with the C7, T1or T2 articular pillar bilaterally.
  Arms: Group 1 Bridge technique mobilization with movement
Other: Dry Needling — Participants in this group received two sessions per week of D.N. treatment for the trapezius muscle.
  Arms: Group 2 Dry Needling

SUMMARY:
This study investigates the effect of the Bridge technique mobilization with movement compared to the Trapezius Dry Needling technique on physiotherapy outcome in patients with cervical dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (25 - 65) years, males & females.
* Cervical dysfunction
* Orthopedic dysfunction without neurological defects
* Limitation in ROM (extension & rotation)
* VAS scale scores for neck pain must be > 4/10
* Neck pain aggravated by neck posture or movement
* Willing to give an informed consent

Exclusion Criteria:

* Any known medical condition, cardio, cancer
* Manipulative treatment within the past three months
* Previous spinal surgery in the past five years
* Current use of medication
* Disc prolapse acute stage
* previous epidural injection since the onset of present symptoms
* diagnosis of any generalized neurological disorder
* medical red flags suggestive of severe pathology
* pregnancy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Numeric Visual analogue scale (VAS) | pre and 1 day post treatment
  Is the most commonly used method for assessing pain intensity. The leftmost value on the 10-cm horizontal line used for VAS indicates a painless condition represented by 0. The rightmost value is 10, which represents extreme pain. The subjects rated their feelings of pain on the line by themselves, thereby quantifying the pain. The validity and reliability are very high.
Quality of life Questionnaire (QoL) | pre and 1 day post treatment
  Is an instrument for measuring the Quality of an individual's life across a broad range of specific areas.
  Quality of life (QoL) could be viewed as a subjective, multidimensional concept that emphasizes an individual's current state's self-perception. However, the general Quality of life includes individuals' evaluation of all aspects of life, including the safety of the environment in which they live, whether they feel they have access to health care and social services, and their current spiritual status
The Northwick Park Neck Pain Questionnaire (NPQ) | pre and 1 day post treatment
  Measures neck pain and consequent patient disabilities. It is easy to complete, to score, and it gives an objective measure to assess the monitor symptoms and outcome in patients with acute or chronic neck pain over time.
Neck Disability Index (NDI) | pre and 1 day post treatment
  The Neck Disability Index (NDI) was grown in (1989) by Howard Vernon. The Index developed to modify the Oswestry Low Back Pain Disability Index with the original author's permission J. Fairbank, (1980). Vernon and Mior at (1991) the reliability and validity analysis finding have been published in the Manipulative and Physiologic Therapeutics Journal.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Quds University, Bethlehem, Palestine, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No